CLINICAL TRIAL: NCT03705039
Title: Assessing the Effects of Pulsed Ultrasound Treatment on Pain, Functionality, Synovial Fluid and Cartilage Thickness, in Knee Osteoarthritis
Brief Title: Is Pulsed Ultrasound Treatment Effective in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Banu Dilek, Principal investigator, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DorkuzEUAli
Record Dates: First submitted 2018-09-24; First posted 2018-10-15 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-03

CONDITIONS: Knee Osteoarthritis
Keywords: knee osteoarthritis; ultrasonography; ultrasound treatment
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: randomized controlled study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Active Comparator): pulsed ultrasound treatment
  Interventions: Other: Pulsed Ultrasound Treatment
- Control Group (Placebo Comparator): sham ultrasound treatment
  Interventions: Other: Control group

INTERVENTIONS:
Other: Pulsed Ultrasound Treatment — Patients will receive treatment with 1 MHz probe with the intensity of 1w/cm2, pulsed at a ratio of 1:4 for 10 minutes and at an interval of 3 sessions per week during 8 weeks, a total of 24 sessions.
  Arms: Treatment Group
Other: Control group — Sham US will be applied to control group for the same times and periods as treatment group. A home exercise program will be given to both of two groups which contains knee range of motion and isometric strengthening exercises.
  Arms: Control Group

SUMMARY:
Osteoarthritis is a progressive rheumatic disease which is the most common cause of musculoskeletal pain and functional impairment, particularly in the elderly group. The most common form is knee osteoarthritis. Pharmacological, non-pharmacological and if required surgical treatment may be applied in the osteoarthritis treatment. Non-pharmacological treatment includes patient education, joint protective measures, exercise, psychological support, diet, weight loss, physical therapy modalities, use of assistive device, hydrotherapy and balneotherapy. Ultrasound therapy is one of the most commonly used physical modalities in osteoarthritis treatment. İt has a deep heating effect and increases tissue regeneration, blood flow and metabolic effects while reducing the inflammation and relaxing the muscles. İn addition, it increases the cartilage regeneration according to certain in vivo and in vitro studies.

Decelerating the cartilage loss and decreasing the high volume of synovial fluid in early-stage knee osteoarthritis is important to preventing progression of the disease. Although there are some randomised controlled clinical trials that prove the effect of ultrasound treatment on pain and functionality in the knee osteoarthritis, there is no study that proves the effect of ultrasound treatment on cartilage thickness and synovial fluid amount. The aim of this study is evaluating the effect of pulsed ultrasound treatment on cartilage regeneration, inflammation and quality of life in the volunteers diagnosed knee osteoarthritis. This study is unique because it is the first study that evaluates the effect of therapeutic pulsed ultrasound on synovial fluid and cartilage thickness with ultrasonography.

DETAILED DESCRIPTION:
The study is a randomised, controlled and parallel group study. 96 patients will be included to study who apply to Dokuz Eylül University Faculty of Medicine, Department of Physical Medicine and Rehabilitation Clinic with the complaint of knee pain, aged between 45-75 years. Patients also have diagnosed as knee osteoarthritis according to American College of Rheumatology (ACR) diagnostic criteria and Kellgren-Lawrence grades are ≤3. These patients will be divided into two groups randomly (Treatment group n:48, control group n:48). The patients in the treatment group will receive treatment with 1 MHz probe with the intensity of 1w/cm2, pulsed at a ratio of 1:4 for 10 minutes and at an interval of 3 sessions per week for 8 weeks, a total of 24 sessions. On the other hand, sham US will be applied to control group for the same times and periods as the treatment group. A home exercise program will be given to both of two groups which contain knee range of motion and isometric strengthening exercises. The patients will be allowed to take paracetamol only when they complain of pain. All patients will be evaluated for 3 times, before and after treatment and 3 months after the treatment with ultrasonographic measurements and life quality tests. Primary aim of this study is to evaluate the effect of pulsed ultrasound on amount of synovial fluid and cartilage thickness.

For this purpose, cartilage thickness and reduction in the amount of synovial fluid will be measured via ultrasound.

Secondary aim is evaluating the effect of pulsed ultrasound on quality of life. Knee pain will be measured by VAS (Visual analogue scale) and functionality will be measured by WOMAC survey and Timed Up and Go Test.

ELIGIBILITY:
Inclusion Criteria:

* Complain of knee pain
* Aged between 45-75 years
* Diagnosed as knee osteoarthritis according to American College of Rheumatology (ACR) diagnostic criteria and Kellgren-Lawrence grades are ≤3

Exclusion Criteria:

* Infection
* Arthritis
* Using corticosteroids
* Corticosteroid injections
* Neurological deficit
* History of knee surgery
* Central and peripheral nerve diseases
* Pregnancy
* Malignancy

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
Amount of synovial fluid | Change from Baseline Amount of synovial fluid at 12 weeks
  The amount of synovial fluid will be measured via ultrasonography in knee

SECONDARY OUTCOMES:
Knee Pain: VAS | All patients will be evaluated for 3 times, at baseline and week 8 and week 12.
  Knee pain will be assessed with Visual Analog Scale (VAS 0-10 cm). Higher values will consider to be worse outcome.
Function | All patients will be evaluated for 3 times at baseline and week 8 and week 12
  Functionally will be assessed with Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) . WOMAC subscores for pain, joint stiffness and daily living activities were calculated separately with likert scale (1 (best) -5 (worst)). Higher values will consider to be worse outcome.
time up and go | All patients will be evaluated for 3 times at baseline and week 8 and week 12
  Functionally will be assessed with time up and go. 3 meters. The patient starts in a seated position.The patient stands up upon therapist's command walks 3 meters, turns around, walks back to the chair and sits down.The time stops when the patient is seated.Higher values will consider to be worse outcome
cartilage thickness in knee | All patients will be evaluated for 3 times at baseline and week 8 and week 12
  cartilage thickness will be measured via ultrasonography in knee

CONTACTS AND LOCATIONS:
Overall Officials: Banu Dilek, MD, Principal Investigator — Dokuz Eylul University
Locations (1):
- Dokuz Eylul University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No